CLINICAL TRIAL: NCT02593955
Title: The Effects of a High Intensity Exercise Training Program on Sleep and Vigilance in Patients With Parkinson's Disease (The Effect of Low Frequency STN DBS on Sleep and Vigilance in PD Patients)
Brief Title: The Effects of a High Intensity Exercise Training Program in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Amy Amara, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F150612003; 5K23NS080912 (NIH)
Record Dates: First submitted 2015-10-28; First posted 2015-11-02 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD exercise group (Active Comparator): Supervised exercise training, 3x per week for 16 weeks
  Interventions: Behavioral: PD exercise
- PD sleep hygeine group (Active Comparator): Tips for improved sleep hygiene, reading materials
  Interventions: Behavioral: Sleep Hygiene
- Healthy control (No Intervention): MRI sub-study only

INTERVENTIONS:
Behavioral: PD exercise — Supervised high intensity exercise 3x/week for 16 weeks
  Arms: PD exercise group
Behavioral: Sleep Hygiene — Sleep medicine physician will provide discuss sleep habits with participants, provide tips for improving sleep hygiene, and provide reading materials.
  Arms: PD sleep hygeine group

SUMMARY:
The purpose of this randomized, controlled interventional study is to determine the effects of a high intensity exercise training program on objective sleep measures, daytime sleepiness, mobility, and brain health/functional connectivity in patients with Parkinson's disease.

DETAILED DESCRIPTION:
The primary outcome measure is the change in sleep efficiency (the number of minutes asleep divided by the number of minutes in bed), as measured by polysomnography. In addition, because patients with Parkinson's disease have excessive sleepiness/impaired vigilance (alertness) and impaired motor function, and because these might be expected to improve with the exercise intervention, this study will also assess vigilance and motor outcomes.

ELIGIBILITY:
Inclusion Criteria: PD participants

1. Subjects with a clinical diagnosis of idiopathic Parkinson's disease based on the presence of bradykinesia and one or both of the following: rest tremor and/or rigidity
2. Hoehn and Yahr stage 2 or 3
3. Stable dopaminergic medication regimen for at least 4 weeks prior to study entry without anticipation of medication change for the duration of the study.
4. Stable doses of medications known to affect sleep and medications for Parkinson's disease for at least 4 weeks prior to study entry without anticipation of medication change for the duration of the study.
5. Age 45 or greater at time of study entry
6. Asymmetric onset of PD
7. Progressive motor symptoms of PD
8. Poor sleep quality (Pittsburgh Sleep Quality Index score >5)
9. MoCA score 18-26
10. Ability to travel to UAB 3x/week for the 16 weeks duration of the study for exercise training sessions as well as for other study visits
11. Subjects must pass a physical examination and PAR-Q to assess exercise readiness

Inclusion Criteria: Healthy Controls

1. Age 45 or greater at time of study entry
2. Poor sleep quality (Pittsburgh Sleep Quality Index score >5)
3. Normal cognition

Exclusion Criteria: PD Participants

1. Atypical features indicative of a Parkinson's Plus disorder (Progressive Supranuclear Palsy, Multiple Systems Atrophy, Corticobasal Degeneration) including cerebellar signs, supranuclear gaze palsy, apraxia, prominent autonomic failure, or other cortical signs.
2. Neuroleptic treatment at time of onset of Parkinsonism
3. Active treatment with a neuroleptic at time of study entry
4. History of multiple strokes with stepwise progression of Parkinsonism
5. History of multiple head injuries
6. Inability to walk without assistance, including a cane, wheelchair, or walker
7. Regular participation in an exercise program within the past 6 months
8. Deep Brain Stimulation
9. Untreated sleep apnea
10. Known narcolepsy
11. Participation in drug studies or the use of investigational drugs within 30 days prior to screening
12. Acute illness or active, confounding medical, neurological, or musculoskeletal conditions that, at the discretion of the PI, would prevent the subject's ability to participate in the study
13. Known contraindication to testing
14. Active alcoholism or other drug addiction
15. Pregnancy

Exclusion criteria for PD subjects undergoing imaging studies:

1. Pacemaker or other metallic object that would make MR imaging unsafe
2. Claustrophobia that prevents participation in imaging portion
3. Any motor, cognitive, or health disorder that in the opinion of the PI would prevent the subject from participating in the imaging portion

Exclusion criteria for healthy controls:

1. Pacemaker or other metallic object that would make MR imaging unsafe
2. Claustrophobia that prevents participation in imaging portion
3. Any motor, cognitive, or health disorder that in the opinion of the PI would prevent the subject from participating in the imaging portion

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in sleep efficiency measured by polysomnography | baseline, week 18, and week 34
  polysomnography
Vigilance outcome measured by psychomotor vigilance task (PVT) | baseline, week 18, and week 34
  psychomotor vigilance task (PVT)
Motor outcome measured by Timed up and go test (TUG) | baseline, week 18, and week 34
  Timed up and go test (TUG)

SECONDARY OUTCOMES:
Home sleep environment | baseline, week 18 and week 34
  comparison of sleep diaries and actigraph related to home sleep environment
MRI Sub-study | baseline (both PD and control), week 18 (PD only)
  comparison of PD and control imaging scans

CONTACTS AND LOCATIONS:
Overall Officials: Amy Amara, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886